CLINICAL TRIAL: NCT01280812
Title: Applying Mobile Persuasive Technologies to Increase Physical Activity in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P0031274; 5R01HL104147-02 (NIH)
Record Dates: First submitted 2010-11-23; First posted 2011-01-21 (Estimated); Results first posted 2020-09-23 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Sedentary Lifestyle; Physical Activity
Keywords: mobile phone; physical activity; women; maintenance; health promotion; prevention
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Maintenance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PA intervention and Maintenance plus (Experimental): 3-month physical activity intervention and 6-month maintenance intervention-Plus program
  Interventions: Behavioral: Mobile phone based physical activity intervention with maintenance plus
- PA intervention and Maintenance regular (Experimental): 3-month physical activity intervention and 6-month maintenance - Regular program
  Interventions: Behavioral: Mobile phone based physical activity intervention with maintenance regular
- Pedometer (Active Comparator): Non-intervention group
  Interventions: Behavioral: Control (pedometer only)

INTERVENTIONS:
Behavioral: Mobile phone based physical activity intervention with maintenance plus — This group will receive a mobile phone software program and a pedometer. Over a 3-month period, participants in this group will be asked to wear a pedometer, use a mobile phone physical activity diary, and respond daily physical activity messages or video clips. Over a 6-month maintenance period, participants will be asked to continue using a pedometer and a mobile phone physical activity diary.
  Arms: PA intervention and Maintenance plus
Behavioral: Mobile phone based physical activity intervention with maintenance regular — This group will receive a mobile phone software program and a pedometer. Over a 3-month period, participants in this group will be asked to wear a pedometer, use a mobile phone physical activity diary, and respond daily physical activity messages or video clips. Over a 6-month maintenance period, participants will be asked to continue using a pedometer.
  Arms: PA intervention and Maintenance regular
Behavioral: Control (pedometer only) — This group will receive a pedometer. Over a 9-month period, participants in this group will be asked to wear a pedometer.
  Arms: Pedometer

SUMMARY:
The primary purpose of this study is to assess the efficacy of the mobile phone-based physical activity intervention on increasing physical activity compared to the control group.

DETAILED DESCRIPTION:
Physical inactivity is associated with increased risk of co-morbidity and premature mortality. Given the rapid growth of mobile phone technology and the increasing number of users, the investigators developed an interactive mobile phone-based physical activity intervention for sedentary women. The investigators propose to conduct a randomized, controlled trial to assess the efficacy of the mobile phone-based physical activity intervention on increasing physical activity over a 3-month period. 192 sedentary women will be randomized in a 2-to-1 ratio to a 3-month mobile phone-based physical activity intervention group or to a control group. To provide insight into how best to maximize the potential for sustained physical activity after completion of the 3-month program, women in the intervention group who complete the physical activity program will be further randomized into a 6-month maintenance intervention-PLUS program (pedometer plus mobile phone diary) or to a 6-month maintenance intervention-REGULAR program (pedometer only). Unlike a conventional maintenance follow-up in which all subjects continue in their respective randomization arms, re-randomizing subjects into either a maintenance intervention-REGULAR group or a maintenance intervention-PLUS group will allow us to examine the "dose-response" of the maintenance methods if the intervention is effective.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle at work and/or during leisure time
* Intend to be physically active
* Female, age >25 to 69
* Access to a home telephone or a mobile phone
* Speak and read English

Exclusion Criteria:

* Known medical conditions or other physical problems that need special attention in an exercise program
* Plan a trip abroad during the first 4 months of the study period.
* Pregnant/Delivered a baby during the last 6 months
* Known severe hearing or speech problem
* Body Mass Index (BMI) > 43.0 kg/m2
* Currently participate in lifestyle modification programs or research studies that may potentially confound the results of the study
* History of bariatric surgery or future plans for bariatric surgery in the next 12 months

Ages: 25 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yoshimi Fukuoka, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California San Francisco (Laurel Heights), San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fukuoka Y, Komatsu J, Suarez L, Vittinghoff E, Haskell W, Noorishad T, Pham K. The mPED randomized controlled clinical trial: applying mobile persuasive technologies to increase physical activity in sedentary women protocol. BMC Public Health. 2011 Dec 14;11:933. doi: 10.1186/1471-2458-11-933. PMID 22168267
- [Background] Fukuoka Y, Gay C, Haskell W, Arai S, Vittinghoff E. Identifying Factors Associated With Dropout During Prerandomization Run-in Period From an mHealth Physical Activity Education Study: The mPED Trial. JMIR Mhealth Uhealth. 2015 Apr 13;3(2):e34. doi: 10.2196/mhealth.3928. PMID 25872754
- [Background] Fukuoka Y, Haskell W, Vittinghoff E. New insights into discrepancies between self-reported and accelerometer-measured moderate to vigorous physical activity among women - the mPED trial. BMC Public Health. 2016 Aug 11;16(1):761. doi: 10.1186/s12889-016-3348-7. PMID 27514368
- [Derived] Lindgren T, Hooper J, Fukuoka Y. Perceptions and Experiences of Women Participating in a Digital Technology-Based Physical Activity Intervention (the mPED Trial): Qualitative Study. JMIR Public Health Surveill. 2019 Dec 20;5(4):e13570. doi: 10.2196/13570. PMID 31859677
- [Derived] Zhou M, Fukuoka Y, Goldberg K, Vittinghoff E, Aswani A. Applying machine learning to predict future adherence to physical activity programs. BMC Med Inform Decis Mak. 2019 Aug 22;19(1):169. doi: 10.1186/s12911-019-0890-0. PMID 31438926
- [Derived] Fukuoka Y, Haskell W, Lin F, Vittinghoff E. Short- and Long-term Effects of a Mobile Phone App in Conjunction With Brief In-Person Counseling on Physical Activity Among Physically Inactive Women: The mPED Randomized Clinical Trial. JAMA Netw Open. 2019 May 3;2(5):e194281. doi: 10.1001/jamanetworkopen.2019.4281. PMID 31125101
- [Derived] Fukuoka Y, Lindgren TG, Mintz YD, Hooper J, Aswani A. Applying Natural Language Processing to Understand Motivational Profiles for Maintaining Physical Activity After a Mobile App and Accelerometer-Based Intervention: The mPED Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jun 20;6(6):e10042. doi: 10.2196/10042. PMID 29925491
- [Derived] Fukuoka Y, Zhou M, Vittinghoff E, Haskell W, Goldberg K, Aswani A. Objectively Measured Baseline Physical Activity Patterns in Women in the mPED Trial: Cluster Analysis. JMIR Public Health Surveill. 2018 Feb 1;4(1):e10. doi: 10.2196/publichealth.9138. PMID 29391341
- [Derived] Fukuoka Y, Lisha NE, Vittinghoff E. Comparing Asian American Women's Knowledge, Self-Efficacy, and Perceived Risk of Heart Attack to Other Racial and Ethnic Groups: The mPED Trial. J Womens Health (Larchmt). 2017 Sep;26(9):1012-1019. doi: 10.1089/jwh.2016.6156. Epub 2017 Apr 18. PMID 28418750

RESULTS

PARTICIPANT FLOW:
Groups:
- Pedometer: Non-intervention group
  Pedometer only: This group will receive a pedometer. Over a 9-month period, participants in this group will be asked to wear a pedometer.
Period: Overall Study
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Pedometer
Started | 70 | 71 | 69
Completed | 67 | 69 | 68
Not Completed | 3 | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Pedometer | Total
Number analyzed (Participants) | 70 | 71 | 69 | 210
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 61 | 65 | 186
  >=65 years | 10 | 10 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (11.2) | 53.6 (11.7) | 51.7 (10.1) | 52.4 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 71 | 69 | 210
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 3 | 13
  Not Hispanic or Latino | 64 | 67 | 66 | 197
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 14 | 14 | 13 | 41
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 9 | 17
  White | 48 | 46 | 38 | 132
  More than one race | 4 | 7 | 9 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 70 | 71 | 69 | 210

OUTCOME MEASURES:

1. Primary Outcome: Accelerometer (Omron Active Style Pro HJA-350IT) Measured Daily Steps
Description: This Omron Active Style Pro HJA-350IT comes with a Universal Serial Bus (USB) Connection and personal computer (PC) Software. The Active Style Pro HJA-350IT can display daily steps. The advantage of using the Omron Active Style Pro HJA-350IT is that the Omron Active Style Pro HJA-350IT will automatically reset the step count every evening at midnight while still allowing participants to view the past 7 days of step counts. Another advantage of using this Omron Active Style Pro HJA-350IT is that a researcher can select 1 of 4 Omron Active Style Pro HJA-350IT screen displays: (1) Steps display only, (2) metabolic equivalents (MET) display only, (3) 24-hour clock display (does not show any physical activity information), and (4) Steps, MET, and weekly average activities during the last four weeks. Data from the most recent 150 days performance will also be automatically stored so they can be directly downloaded to a computer.
Time Frame: Baseline, 3, and 9 months
Population: Intention to treat (ITT) analysis
Measure: Mean (Standard Deviation); unit: Steps/Day
Groups:
- Control: Non-intervention group
  Pedometer only: This group will receive a pedometer. Over a 9-month period, participants in this group will be asked to wear a pedometer.
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
Number analyzed (Participants) | 70 | 71 | 69
Steps/Day
  Mean total daily steps at baseline | 5837 (3235) | 5063 (2526) | 5384 (2920)
  Mean total daily steps at 3 months | 8709 (3910) | 8096 (3903) | 6608 (3719)
  Mean total daily steps at 9 months | 7807 (4093) | 6909 (3704) | 6265 (3524)
Statistical Analysis 1: Comparison: PA Intervention and Maintenance Plus vs PA Intervention and Maintenance Regular vs Control; Intent to treat analysis; Test type: Superiority; Mixed Models Analysis; Two-sided P values less than .05 were considered statistically significant; Median Difference (Net) = 1100, Standard Deviation 3000

2. Primary Outcome: Accelerometer (Omron Active Style Pro HJA-350IT) Measured Moderate to Vigorous Physical Activity (Minutes Per Day)
Description: as for outcome 1
Time Frame: Baseline, 3 and 9 months
Population: Intention to treat (ITT) analysis
Measure: Mean (Standard Deviation); unit: minutes per day
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Pedometer
Number analyzed (Participants) | 70 | 71 | 69
minutes per day
  Mean Daily MVPA at baseline | 43.5 (29.6) | 38.0 (24.4) | 45.7 (33.4)
  Mean Daily MVPA at 3 months | 67.6 (34.9) | 61.6 (33.3) | 53.0 (38.0)
  Mean Daily MVPA at 9 months | 60.1 (33.7) | 56.6 (36.4) | 50.8 (34.4)

3. Secondary Outcome: Self-reported Physical Activity Measured by the 7-day Physical Activity Recall (PAR)
Description: An interviewer-administered 7-day physical activity recall (PAR) is used to assess physical activities performed during the week preceding each visit. The PAR is a widely used and well-validated self-report recall instrument that assesses the frequency, duration, and intensity of physical activity. It yields average kcal/kg/day.
Time Frame: Baseline, 3 and 9 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: kcal/kg/day
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
Number analyzed (Participants) | 70 | 71 | 69
kcal/kg/day
  kcal/kg/day at baseline | 33.1 (1.07) | 32.9 (1.09) | 32.9 (1.42)
  kcal/kg/day at 3 months | 34.5 (1.75) | 34.8 (2.14) | 33.7 (1.78)
  kcal/kg/day at 9 months | 34.3 (2.22) | 33.8 (1.90) | 34.1 (2.69)

4. Secondary Outcome: Modified Self-Efficacy for Physical Activity Survey
Description: The Self-Efficacy for Physical Activity will be used to measure how confident the participant is to engage in physical activity in a specific situation. A sample item is, "I am confident I can participate in regular physical activity when I am tired." The measure consists of five items on a scale of 1 to 5, "1" being "not at all confident" and "5" being "very confident." The possible range of scores is from 5 to 25 points. Higher scores indicate higher self-efficacy for physical activity. Reported internal consistency ranges from 0.78 to 0.82. This measure has been widely used in adult women and men. Based on our pilot study, we added one additional question to this survey.
Time Frame: Baseline, 3 and 9 months
Population: Intent to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
Number analyzed (Participants) | 70 | 71 | 69
units on a scale
  Self-efficacy at baseline | 19.0 (4.79) | 19.8 (5.09) | 18.8 (3.95)
  Self-efficacy at 3 months | 18.1 (4.50) | 18.0 (5.13) | 19.1 (5.53)
  Self-efficacy at 9 months | 18.3 (4.93) | 17.8 (5.24) | 19.2 (5.13)

5. Secondary Outcome: Social Support for Physical Activity (Family)
Description: The Social Support and Exercise Survey will be used to measure both friend and family social support related to physical activity during the past three months. The measure comprises two subscales (friend and family support subscales). Each subscale has 12 items with 5-point Likert scales (ranging from 1, "none" to 5, "very often"). The ratings of all 12 items are summed for a subtotal score (possible ranges from 12 to 60). Internal consistency (Cronbach's alpha) of the measure was 0.83 in previous studies. Test-retest reliabilities of the measure have ranged from 0.79 to 0.90 for both scales. Reported internal consistencies ranged between 0.80 to 0.93 for both scales. Higher scores indicate greater support.
Time Frame: Baseline, 3 and 9 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
Number analyzed (Participants) | 70 | 71 | 69
units on a scale
  Physical activity social support from family at baseline | 32.8 (9.16) | 31.5 (10.9) | 32.0 (9.18)
  Physical activity social support from family at 3 months | 34.8 (10.7) | 35.6 (11.2) | 31.6 (9.94)
  Physical activity social support from family at 9 months | 34.3 (11.1) | 34.5 (9.86) | 33.4 (11.0)

6. Secondary Outcome: Social Support for Physical Activity (Friends)
Description: The Social Support and Exercise Survey will be used to measure both friend and family social support related to physical activity during the past three months. The measure comprises two subscales (friend and family support subscales). Each subscale has 12 items with 5-point Likert scales (ranging from 1, "none" to 5, "very often"). The ratings of all 12 items are summed for a subtotal score (possible ranges from 12 to 60). Internal consistency (Cronbach's alpha) of the measure was 0.83 in previous studies. Test-retest reliabilities of the measure have ranged from 0.79 to 0.90 for both scales. Reported internal consistencies ranged between 0.80 to 0.93 for both scales.
Time Frame: Baseline, 3 and 9 months
Population: Intention to treat analysis
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
Number analyzed (Participants) | 70 | 71 | 69
units on a scale
  PA social support from friend at baseline | 31.8 (8.11) | 31.5 (8.21) | 31.1 (8.91)
  PA social support from friend at 3 months | 34.7 (8.36) | 35.1 (8.48) | 31.1 (8.35)
  PA social support from friend at 9 months | 35.4 (9.17) | 33.9 (9.17) | 31.8 (8.74)

ADVERSE EVENTS:
Time Frame: 9 months in total: -Intervention (Plus and Regular Groups) versus Control Group during the 3-month intervention period and the 6-month maintenance period.
Groups:
- PA Intervention and Maintenance Regular: 3-month physical activity intervention and 6-month maintenance intervention regular program
  Over a 3-month period, participants in this group will be asked to wear a pedometer, use a mobile phone physical activity diary, and respond daily physical activity messages or video clips. Over a 6-month maintenance period, participants will be asked to stop using the app (activity diary).
Arm/Group | PA Intervention and Maintenance Plus | PA Intervention and Maintenance Regular | Control
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/71 | 0/69
Serious Adverse Events (participants affected / at risk) | 1/70 | 1/71 | 3/69
Other Adverse Events (participants affected / at risk) | 11/70 | 10/71 | 6/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Intervention and Maintenance Plus (N=70) | PA Intervention and Maintenance Regular (N=71) | Control (N=69)
Hospitalization (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Hospitalization (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hospitalization (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hospitalization (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PA Intervention and Maintenance Plus (N=70) | PA Intervention and Maintenance Regular (N=71) | Control (N=69)
Emergency Department or Urgent Care Facility Visit (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0)
Emergency Department or Urgent Care Facility Visit (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Emergency Department or Urgent Care Facility Visit (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3)
Emergency Department or Urgent Care Facility Visit (Injury, poisoning and procedural complications) | 3 (4) | 3 (3) | 0 (0) — car accident, assault, head injury at work, burn
Emergency Department or Urgent Care Facility Visit (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Emergency Department or Urgent Care Facility Visit (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Emergency Department or Urgent Care Facility Visits (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Emergency Department or Urgent Care Facility Visit (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 1 (1)
Emergency Department or Urgent Care Facility Visit (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Emergency Department or Urgent Care Facility Visit (Investigations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No